CLINICAL TRIAL: NCT03054168
Title: The Regulation of Skeletal Muscle Protein Synthesis by Systemic Hormones and Its Influence on Ageing and Anabolic Resistance
Brief Title: Systemic Hormones and Muscle Protein Synthesis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Philip Atherton, Philip Atherton, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Hormones
Record Dates: First submitted 2017-02-10; First posted 2017-02-15 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Sarcopenia; Muscle Hypotrophy; Muscle Atrophy
Keywords: Protein Synthesis; Hypertrophy; Testosterone
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy; Hypertrophy | interventions — Testosterone; Goserelin; Gonadotropin-Releasing Hormone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: To achieve our aims we will recruit 16 young healthy males (Age: 18-30 y; BMI: 18-30kg/m2) and 16 older healthy males (Age: 65-75 y; BMI: 18-30kg/m2). Volunteers will then be randomly assigned to a testing group; 1) Young placebo trained (N=10), 2) Young gonadotropin releasing hormone analogue trained (3.6mg Zoladex subcutaneous injection (every 4 weeks) N=10), 3) Old placebo trained (N=10) and 4) Old Testosterone trained (Sustanon 250: 250 mg every 2-3wks intramuscular injection, N=10). All participants will receive whole body resistance exercise training for six weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Old Testosterone trained (Experimental): 8 old participants (65-75 years old) who will receive resistance exercise training and Testosterone (Sustanon 250: 250 mg every 2wks)
  Drug name: Sustanon 250 Generic Name: Testosterone Proprietary Name: N/A Formulation: 250mg of Testosterone in 1ml volume Dose: 250mg of testosterone Frequency: every 2 weeks Route: intramuscular injection
  Interventions: Drug: Sustanon 250
- Old Placebo trained (Placebo Comparator): 8 old participants (65-75 years old) who will receive resistance exercise training and Placebo every two weeks.
  Interventions: Other: Placebo
- Young Zoladex trained (Experimental): 8 young participants (18-30 years old) who will receive resistance exercise training and Testosterone inhibitor (3.6mg Zoladex subcutaneous injection, one time over the study)
  Drug name: Zoladex Generic Name: Gonadotropin-releasing hormone analogue; Goserelin Proprietary Name: N/A Formulation: Solution for injection Dose: 3.6mg Frequency: Single injection one time over the study. Route: Subcutaneous injection (abdomen) performed by clinician.
  Interventions: Drug: Zoladex
- Young placebo trained (Placebo Comparator): 8 young participants (18-30 years old) who will receive resistance exercise training and placebo, one time over the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sustanon 250 — The frequency of the injection will be every 2 weeks, 250mg of testosterone, intramuscular injection.
  Other Names: Testosterone
  Arms: Old Testosterone trained
Drug: Zoladex — The frequency of the injection will be just one injection, 3.6 mg of Zoladex, Subcutaneous injection (abdomen).
  Other Names: Gonadotropin-releasing hormone analogue; Goserelin
  Arms: Young Zoladex trained
Other: Placebo
  Other Names: Saline
  Arms: Old Placebo trained; Young placebo trained

SUMMARY:
This study evaluates the effect of increase in testosterone levels in older males and the effects of decrease in testosterone levels in young males on muscle protein synthesis.

DETAILED DESCRIPTION:
Skeletal muscle represents the largest organ in the body, comprising >50% of total body mass. The function of skeletal muscle is best understood for its role in locomotion and providing mechanical support to the skeleton to facilitate movement. However, skeletal muscles are also important for maintaining whole-body metabolic health. For example, muscles also act as a site for glucose disposal thereby acting to maintain whole-body glycaemic control. In addition, skeletal muscles represent a vast protein store, the amino acids from which can be used in times of fasting, infection and disease to provide energy to maintain other critical organs. Exercise (resistance type exercise (RE-T) in particular) still remains the most effective means by which to maintain and increase muscle mass through stimulation of muscle protein synthesis (MPS), despite this, how exercise regulates these changes in muscle mass is still unknown. A number of pathways have been inferred as key, however it is clear from a number of studies that systemic hormone levels, testosterone in particular, may provide a significant contribution. It is well known that chronic androgenic hormone deficiency can lead to a loss of lean body mass and strength, which can in turn contribute to impaired physical function. Furthermore, when testosterone levels are pharmacologically reduced (using a gonadotropin releasing hormone analogue) in healthy young males, resistance exercise training induced increases in muscle mass and strength are absent. Whilst systemic hormone levels are carefully maintained in youth (unless illness or deficiency is present), levels of these hormones decrease with age, particularly in those that are not regularly physically active, indeed approximately 25-30% of older men have levels of testosterone which are below the threshold used to define hypogonadism. Therefore, there is significant need to understand the underlying mechanisms behind hormonally induced muscle mass regulation. Furthermore, in older age there is a resistance to traditional anabolic stimuli such as nutrition or resistance exercise, with older adults showing a blunted-anabolic hormonal profile in response to resistance training compared to young. These impairments to hormonal regulation with ageing may in part be responsible for the slow decline in muscle mass with age known as sarcopenia. Whilst all muscle-wasting conditions are of considerable concern, it is the loss of muscle in older age that poses the greatest socio-economic burden. Therefore there is a significant clinical need to identify contributing factors to this muscle loss so that they can be specifically targeted for intervention (i.e., pharmacological hormonal therapies).

The aims of this project are two fold: 1) Firstly we aim to investigate the impact of systemic hormone levels on control of muscle mass in healthy young adults undertaking a resistance exercise training program, we hypothesize that reduction of hormone levels in systemically normal young adults will impair MPS and muscle mass gains in response to resistance exercise training. 2) Secondly we aim to investigate the impact of enhancing testosterone levels in older adults on responsiveness to resistance exercise training and the contribution of systemic testosterone levels to muscle mass regulation in ageing, we hypothesize that increasing testosterone levels in older males will improve responsiveness to anabolic stimuli (RE-T).

ELIGIBILITY:
Inclusion Criteria:

Young (18-30y) and old (60-75y) males who are generally healthy

Exclusion Criteria:

* Participation in a formal exercise regime
* BMI < 18 or > 30 kg·m2
* Active cardiovascular disease:

  * uncontrolled hypertension (BP > 160/100),
  * angina,
  * heart failure (class III/IV),
  * arrhythmia,
  * right to left cardiac shunt,
  * recent cardiac event
* Taking beta-adrenergic blocking agents, statins, non-steroidal anti-inflammatory drugs or HRT
* Cerebrovascular disease:

  * previous stroke,
  * aneurysm (large vessel or intracranial)
  * epilepsy
* Respiratory disease including:

  * pulmonary hypertension,
  * COPD,
  * asthma,
* Metabolic disease:

  * hyper and hypo parathyroidism,
  * Hypo and hyper gonadism
  * untreated hyper and hypothyroidism,
  * Cushing's disease,
  * type 1 or 2 diabetes
* Active inflammatory bowel or renal disease
* Malignancy
* Altered hormonal profile
* Recent steroid treatment (within 6 months) or hormone replacement therapy
* Clotting dysfunction
* Musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants are male.
Enrollment: 34 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2019-02-15 (Estimated)

PRIMARY OUTCOMES:
Muscle Protein Synthesis | 0-6 Weeks
  Comparison of muscle protein synthesis between young and older individuals when their testosterone levels decrease and increase, respectively; in response to 6 weeks whole body resistance exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Atherton, Professor, Principal Investigator — The University of Nottingham; Nathaniel Szewczyk, Ass. Proff, Study Chair — The University of Nottingham
Locations (1):
- Royal Derby Hospital Medical School, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mauras N, Hayes V, Welch S, Rini A, Helgeson K, Dokler M, Veldhuis JD, Urban RJ. Testosterone deficiency in young men: marked alterations in whole body protein kinetics, strength, and adiposity. J Clin Endocrinol Metab. 1998 Jun;83(6):1886-92. doi: 10.1210/jcem.83.6.4892. PMID 9626114
- [Background] Kvorning T, Andersen M, Brixen K, Madsen K. Suppression of endogenous testosterone production attenuates the response to strength training: a randomized, placebo-controlled, and blinded intervention study. Am J Physiol Endocrinol Metab. 2006 Dec;291(6):E1325-32. doi: 10.1152/ajpendo.00143.2006. Epub 2006 Jul 25. PMID 16868226
- [Background] Abbasi AA, Drinka PJ, Mattson DE, Rudman D. Low circulating levels of insulin-like growth factors and testosterone in chronically institutionalized elderly men. J Am Geriatr Soc. 1993 Sep;41(9):975-82. doi: 10.1111/j.1532-5415.1993.tb06764.x. PMID 8409184
- [Background] Harman SM, Metter EJ, Tobin JD, Pearson J, Blackman MR; Baltimore Longitudinal Study of Aging. Longitudinal effects of aging on serum total and free testosterone levels in healthy men. Baltimore Longitudinal Study of Aging. J Clin Endocrinol Metab. 2001 Feb;86(2):724-31. doi: 10.1210/jcem.86.2.7219. PMID 11158037
- [Background] Baker JR, Bemben MG, Anderson MA, Bemben DA. Effects of age on testosterone responses to resistance exercise and musculoskeletal variables in men. J Strength Cond Res. 2006 Nov;20(4):874-81. doi: 10.1519/R-18885.1. PMID 17194250
- [Background] Kumar V, Selby A, Rankin D, Patel R, Atherton P, Hildebrandt W, Williams J, Smith K, Seynnes O, Hiscock N, Rennie MJ. Age-related differences in the dose-response relationship of muscle protein synthesis to resistance exercise in young and old men. J Physiol. 2009 Jan 15;587(1):211-7. doi: 10.1113/jphysiol.2008.164483. Epub 2008 Nov 10. PMID 19001042
- [Background] Vingren JL, Kraemer WJ, Ratamess NA, Anderson JM, Volek JS, Maresh CM. Testosterone physiology in resistance exercise and training: the up-stream regulatory elements. Sports Med. 2010 Dec 1;40(12):1037-53. doi: 10.2165/11536910-000000000-00000. PMID 21058750